CLINICAL TRIAL: NCT04741958
Title: Role of Ultrasound Guided Percutaneous Transthoracic Core Needle Biopsy in Diagnosis of Peripheral Thoracic Tumors
Brief Title: Role of Ultrasound Guided Peripheral Thoracic Tumors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Beni-Suef University (Other)
Responsible Party: Principal Investigator, Maha Fathy, lecturer of chest, Beni-Suef University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: role of us guided in in PTT
Record Dates: First submitted 2020-10-17; First posted 2021-02-05 (Actual); Last update posted 2021-02-05 (Actual); Status verified 2021-02

CONDITIONS: Thoracic Neoplasms
Keywords: Ultrasound; .; Chest; Diseases; Core needle biopsy
MeSH Terms: conditions — Thoracic Neoplasms; Disease

STUDY DESIGN:
Intervention Model Description: The current study is a case series study conducted on 60 patients that had radiographic evidence of thoracic mass suspected of malignancy
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ultra sound guided percutaneous core needle biopsy (Experimental): 60 patients that had radiographic evidence of thoracic mass suspected of malignancy .Twenty masses were in the lung, seventeen lesions were in the pleura, ten masses were in the mediastinum, eleven enlarged palpable lymph nodes, and two masses were in chest wall. The sensitivity, PPV and accuracy for detection of chest tumors in chest wall, mediastinum, lung, and pleura were (100 %) for all, and in LN (88.9, 100 and 90.9 %) respectively. The overall diagnostic performance of sonar guided true cut needle biopsy in diagnosis was 97.78 % sensitivity, 98.18% accuracy, and 100 % PPV
  Interventions: Diagnostic Test: Ultrasound Guided Peripheral Thoracic Tumors

INTERVENTIONS:
Diagnostic Test: Ultrasound Guided Peripheral Thoracic Tumors — Transthoracic ultrasonography: Transthoracic US was done using machine Hitachi 5500 in the Diagnostic Ultrasound Unit - Chest Department- Kasr El-Aini Hospital.on 60 patients that had radiographic evidence of thoracic mass suspected of malignancy

SUMMARY:
The aim of the study was to calculate sensitivity, and accuracy of ultrasound guided percutaneous core needle biopsy in different thoracic tumors (lung, pleural, chest wall and mediastinal).

DETAILED DESCRIPTION:
Peripheral intrathoracic shadows are common presentation of different diseases of different origin (chest wall, pleura, pulmonary, and mediastinum), they are increasing in numbers including, peripheral lung cancer, tuberculosis, pneumonia, and atelectasis. [1] Thoracic masses with wall contact represent a frequent pathology that requires complex imaging studies, and often interventional procedures, in order to reach the complete diagnosis. In most cases, after a thoracic lesion is found on a thoracic X-Ray, the next step is to perform a CT and/or a bronchoscopy exam, but pleural and pulmonary lesions often call for additional investigations.

Therefore, transthoracic ultrasonography (US) permits visualization of these lesions, their structural characterization, while offering suggestive elements for their malignant nature and for the differential diagnosis.

Sonography has the capacity to clarify the nature of opaque lesions such as effusions, atelectasis, masses, and consolidations. Transthoracic ultrasound has received increased interest from chest Physicians in recent years as it has the advantages of bedside availability, absence of radiation, and guided aspiration of fluid-filled areas and solid tumors.

Furthermore US allows percutaneous guided biopsies with lower risks compared with the radiological guiding methods (fluoroscopy and CT). Trransthoracic US can replace other imaging modalities of the chest and guide a variety of diagnostic and therapeutic procedures. Under real time US guidance, the success rate of transthoracic needle aspiration or biopsy (TNB) significantly increases, whereas the risk of complications is greatly reduced.

ELIGIBILITY:
Inclusion Criteria:

1. An acoustic window for the ultrasound beam to penetrate.
2. Patients have platelet count more than 100000 and normal prothrombin time.

Exclusion Criteria:

1. Cardio vascular instability.
2. Arterio venous malformation or aneurysm.
3. Patients with uncontrolled convulsions

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2020-09-12 (Actual); Primary Completion 2020-11-01 (Actual); Study Completion 2020-12-01 (Actual)

PRIMARY OUTCOMES:
Value of sonar guided true cut needle biopsy in diagnosis in different thoracic tumors (lung, pleural, chest wall and mediastinal). | 8week
  diagnostic performance of sonar guided true cut needle biopsy in diagnosis in different thoracic tumors (lung, pleural, chest wall and mediastinal) in 60 patients that had radiographic evidence of thoracic mass suspected of malignancy by measure sensitivity, accuracy, and Positive predictive values
  * True positive result: the tumor is confirmed by a definite histopathologic diagnosis made by Tru-Cut core biopsy
  * True negative result: case not diagnosed as a tumor by ultrasound Tru-Cut core biopsy & this finding was confirmed by another modality for biopsy
  * False negative result was considered to have occurred if the tumor wasn't diagnosed by ultrasound guided biopsy, and the tumor was confirmed using other modalities (CT guided, Thoracoscopic, or surgical biopsy).

CONTACTS AND LOCATIONS:
Overall Officials: maha fathy, MD of chest, Principal Investigator — beni seuf unversity
Locations (1):
- Benisuef Unversity, Banī Suwayf, Egypt

REFERENCES:
- [Result] Rivera MP, Detterbeck F, Mehta AC; American College of Chest Physicians. Diagnosis of lung cancer: the guidelines. Chest. 2003 Jan;123(1 Suppl):129S-136S. doi: 10.1378/chest.123.1_suppl.129s. PMID 12527572
- [Result] Chira R, Chira A, Mircea PA. Intrathoracic tumors in contact with the chest wall--ultrasonographic and computed tomography comparative evaluation. Med Ultrason. 2012 Jun;14(2):115-9. PMID 22675711
- [Result] Balik M, Plasil P, Waldauf P, Pazout J, Fric M, Otahal M, Pachl J. Ultrasound estimation of volume of pleural fluid in mechanically ventilated patients. Intensive Care Med. 2006 Feb;32(2):318. doi: 10.1007/s00134-005-0024-2. Epub 2006 Jan 24. PMID 16432674
- [Result] Diacon AH, Theron J, Schubert P, Brundyn K, Louw M, Wright CA, Bolliger CT. Ultrasound-assisted transthoracic biopsy: fine-needle aspiration or cutting-needle biopsy? Eur Respir J. 2007 Feb;29(2):357-62. doi: 10.1183/09031936.00077706. Epub 2006 Nov 1. PMID 17079257
- [Result] Chira RI, Chira A, Mircea PA, Valean S. Mediastinal masses-transthoracic ultrasonography aspects. Medicine (Baltimore). 2017 Dec;96(49):e9082. doi: 10.1097/MD.0000000000009082. PMID 29245326
- [Result] Hafez MR, Sobh ES, Elsawy SB, Abo-Elkheir OI. The usefulness of thoracic ultrasonography in diagnosis and staging of bronchogenic carcinoma. Ultrasound. 2017 Nov;25(4):200-212. doi: 10.1177/1742271X17721264. Epub 2017 Aug 3. PMID 29163656
- [Result] Schubert P, Wright CA, Louw M, Brundyn K, Theron J, Bolliger CT, Diacon AH. Ultrasound-assisted transthoracic biopsy: cells or sections? Diagn Cytopathol. 2005 Oct;33(4):233-7. doi: 10.1002/dc.20342. PMID 16138366
- [Result] Yang PC, Luh KT, Chang DB, Wu HD, Yu CJ, Kuo SH. Value of sonography in determining the nature of pleural effusion: analysis of 320 cases. AJR Am J Roentgenol. 1992 Jul;159(1):29-33. doi: 10.2214/ajr.159.1.1609716.